CLINICAL TRIAL: NCT01693016
Title: Validation of Non-invasive Hb-measurement (SpHb) in Children With the Masimo@ Radical 7
Brief Title: Validation of Non-invasive Hemoglobin (SpHb) Measurement in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Eva Wittenmeier, Dr. Eva Wittenmeier, Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MASIMO 2012
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Non-invasive Hb Measurement in Children
Keywords: non-invasive Hb measurement in children
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- inhalation group (Other): 20 children Taking blood samples and SpHb-measurement was made under inhalational anesthesia
  Interventions: Device: non-invasive measurement of Hb; Procedure: taking blood samples
- non-inhalational (Other): 40 children Taking blood samples and SpHb measurements in awake and spontaneous breathing children.
  Interventions: Device: non-invasive measurement of Hb; Procedure: taking blood samples

INTERVENTIONS:
Device: non-invasive measurement of Hb
  Other Names: SpHb (®) by Masimo ® Radical 7
Procedure: taking blood samples
  Other Names: blood for BGA (ABL 800); blood for laboratory Hb (Siemens Advia)

SUMMARY:
The purpose of this study is to evaluate the value of the new technique of non-invasive measurement of Hb in children undergoing a surgical procedure.

DETAILED DESCRIPTION:
Several surgical procedures require haemoglobin monitoring due to possible blood loss and the need of blood transfusion. The standard for monitoring hemoglobin (Hb) is the measurement of blood samples. The novel technique of non-invasive continuous measurement of Hb using Pulse CO-Oximetry may allow measuring Hb without obtaining blood samples.

This new technique has not been tested yet in children undergoing anesthesia for elective surgical procedures. In this study the investigators compare the non-invasive Hb measurement with Masimo® technology (SpHb) with the standard Hb measurement using ABL-800 Flex (BGA) and Siemens Advia (labHb, reference method) before the children undergo the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* children (>= 3 kg until 8 years)
* ASA I-III
* written informed consent of legal representative

Exclusion Criteria:

* children <= 3kg or > 8 years
* emergency surgery
* allergy against sensor of SpHb(®)
* artery occlusive disease
* sepsis
* haemoglobinopathy
* specific medical or psychological circumstances which do not allow the consent of the legal representative or the performance of the study

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
correlation between SpHb(®) and the Hb measured by the ABL800Flex and the Siemens Advia | one day

SECONDARY OUTCOMES:
influence of inhalation anesthetics | one day
  The blood samples are taken from the needle infusion set the child gets for anesthesia. Some children will need an inhalational induction of anesthesia before they can get the needle and the sensor for the SpHb (®) monitoring. So an influence of the application of inhalation anesthetics on the accuracy of the SpHb (®) will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Wittenmeier, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Dr. Eva Wittenmeier, Mainz, Germany

REFERENCES:
- [Derived] Wittenmeier E, Bellosevich S, Mauff S, Schmidtmann I, Eli M, Pestel G, Noppens RR. Comparison of the gold standard of hemoglobin measurement with the clinical standard (BGA) and noninvasive hemoglobin measurement (SpHb) in small children: a prospective diagnostic observational study. Paediatr Anaesth. 2015 Oct;25(10):1046-53. doi: 10.1111/pan.12683. Epub 2015 Jul 14. PMID 26179143